CLINICAL TRIAL: NCT04868747
Title: The Effect of Perioperative Lidocaine Intravenous Infusion on Neutrophil Extracellular Trapping After Surgery for Stomach Cancer
Brief Title: The Effect of Perioperative Lidocaine Infusion on Neutrophil Extracellular Trapping
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to financial problem
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NET-lidocaine-stomach cancer
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): The study group receives the intravenous 1% lidocaine 1.5 mg/kg bolus followed by 1.5 mg/kg/h during surgery and 1.0 mg/kg/h until 24 hours after surgery (Max.<120 mg/h).
  Interventions: Drug: Lidocaine
- control group (Placebo Comparator): The control group receives intravenous normal saline 0.15 ml/kg bolus followed by 0.15 ml/kg/h during surgery and 0.1 mg/kg/h until 24 hours after surgery.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Lidocaine — The participants receive perioperative lidocaine infusion with general anesthesia for gastrectomy.
  Arms: study group
Drug: normal saline — The participants receive perioperative normal slaine infusion with general anesthesia for gastrectomy.
  Arms: control group

SUMMARY:
To investigate the effect of perioperative lidocaine infusion on the neutrophil extracellular trapping after minimally invasive surgery for stomach cancer

DETAILED DESCRIPTION:
To investigate the effect of perioperative lidocaine infusion on the neutrophil extracellular trapping, especially citrullinated histone3, neutrophil elastase, myeloperoxidase

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stomach cancer
* ASA class I-III
* no metastatic disease

Exclusion Criteria:

* hepatic, renal disease
* chronic inflammatory disease, eg. rheumatoid arthritis
* steroid or anti-inflammatory drug medication
* allergies to study drugs
* neuropsychiatric disease
* refusal of participation
* breast feeding or pregnancy
* weight < 40 kg

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
serum concentration of NET(neutrophil extracellular trapping)-related biomarker | 24 hours after surgery
  NET-related biomarker (citrullinated histone3, neutrophil elastase, myeloperoxidase)

SECONDARY OUTCOMES:
quality of recovery | 24 hours after surgery
  The quality of recovery is assessed using questionnaire. This questionnaire includes 15 items. The score range is from 0 to 150. The higher score means the better quality of recovery after surgery.
postoperative pain | 24 hours after surgery
  The postoperative pain is assessed using numeric rating scale (NRS; 0=no pain, 10=the maximal pain)
survival of patients | 5 years
  The survival of patients is assessed using electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Young Eun Moon, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea